CLINICAL TRIAL: NCT00386282
Title: Acceptability and Feasibility of Medical Abortion in Mexico, Puerto Rico, Armenia and Azerbaijan: A Study of Buccal Misoprostol Administration Following Mifepristone 200 mg for Abortion up to 63 Days' Gestation
Brief Title: Acceptability and Feasibility of Medical Abortion Using Mifepristone and Buccal Misoprostol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.4
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Abortion, First Trimester
Keywords: Mifepristone; Misoprostol; Buccal administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mifepristone-misoprostol treatment (Other): 200 mg mifepristone followed by 800 mcg buccal misoprostol 24-48 hours after the mifepristone
  Interventions: Drug: mifepristone-misoprostol treatment

INTERVENTIONS:
Drug: mifepristone-misoprostol treatment — 200 mg mifepristone followed by 800 mcg buccal misoprostol 24-48 hours after the mifepristone.
  Other Names: medical abortion

SUMMARY:
This study examined the acceptability and feasibility of introducing a mifepristone-misoprostol regimen of medical abortion into abortion services in two private clinics in Puerto Rico; 2 clinics in Baku, Azerbaijan; 3 clinics in Yerevan, Armenia; and 4 clinics in Mexico City. It was hypothesized that the study regimen would be both acceptable and efficacious.

DETAILED DESCRIPTION:
The study recruited women with pregnancies up to 63 days gestation. Eligible women took 200 mg mifepristone, followed by 800 buccal misoprostol. They later underwent clinic follow-up to determine if their medical abortions were complete. The study assessed the acceptability and feasibility of the above regimen and sought to determine the efficacy and acceptability of buccal administration of misoprostol as well as the acceptability of side effects experienced by women.

ELIGIBILITY:
Inclusion Criteria:

* Gestation up to 63 days
* General good health
* Willingness to provide contact information for follow-up
* Absence of conditions which contraindicate the use of mifepristone and misoprostol for pregnancy termination

Exclusion Criteria:

* Ectopic pregnancy
* Intrauterine device (IUD) in place

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2006-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
efficacy | 15 days

SECONDARY OUTCOMES:
acceptability | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Hector Diaz Martinez, MD, Principal Investigator — Clinica de Planificacion Familiar; Angela Arredondo, MD, Principal Investigator — Woman's Metropolitan Center; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Gulnara Rzaeva, MD, Principal Investigator — Scientific Research Institute of Obstetrics & Gynecology; Besti Muradova, MD, Principal Investigator — Family Planning Center; Susanna Fildjyan, MD, Principal Investigator — Institute of Perinatology, Obstetrics and Gynecology; Armine Harutyunyan, MD, Principal Investigator — Center for Family Planning and Sexual Health; Anna Aghajanyan, MD, Principal Investigator — State Medical University; Ranulfo Rios, MD, Principal Investigator — H G Enrique Cabrera; Laura Garcia Martinez, MD, Principal Investigator — H.M.I Inguaran; Antonio E Flores, MD, Principal Investigator — C S Beatriz Velasco Aleman; Elba Margarita Lugo Hernandez, MD, Principal Investigator — C S Santa Catarina
Locations (11):
- Armenia (3):
  - Center for Family Planning and Sexual Health, Yerevan
  - Institute of Perinatology, Obstetrics and Gynecology, Yerevan
  - State Medical University, Yerevan
- Azerbaijan (2):
  - Family Planning Center, Baku
  - Scientific Research Institute of Obstetrics and Gynecology, Baku
- Mexico (4):
  - C.S. Beatriz Velasco Aleman, Mexico City, Federal District
  - C.S. Santa Catarina, Mexico City, Federal District
  - H.G. Enrique Cabrera, Mexico City, Federal District
  - H.M.I Inguaran, Mexico City, Federal District
- Puerto Rico (2):
  - Clinica de Planificacion Familiar, Lomas Verdes, Bayamon
  - Woman's Metropolitan Center, San Juan

REFERENCES:
- [Derived] Pena M, Dzuba IG, Smith PS, Mendoza LJ, Bousieguez M, Martinez ML, Polanco RR, Villalon AE, Winikoff B. Efficacy and acceptability of a mifepristone-misoprostol combined regimen for early induced abortion among women in Mexico City. Int J Gynaecol Obstet. 2014 Oct;127(1):82-5. doi: 10.1016/j.ijgo.2014.04.012. Epub 2014 Jun 4. PMID 24957534